CLINICAL TRIAL: NCT04003896
Title: A Pilot Study to Evaluate the Response and Tolerability of Verzenio (Abemaciclib) in Patients With Advanced Biliary Tract Carcinoma
Brief Title: A Study to Evaluate Abemaciclib in Advanced Biliary Tract Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The manufacturer and funder Eli Lilly requested to terminate the study
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Nelson Yee, MD, PhD, Associate Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-18-052
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Biliary Tract Carcinoma
Keywords: Biliary Tract Carcinoma; Abemaciclib
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: This is a pilot study to confirm tolerability of abemaciclib and provide an estimate of the overall response rate. A sample size of 10 subjects is determined to be minimally sufficient for these pilot study objectives. There will be no protocol scheduled hiatus and daily dosing will be continuous unless there is unacceptable toxicity, disease progression, or death.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib (Experimental): Abemaciclib will be given as a single oral agent A sample size of 10 subjects is determined to be minimally sufficient for these pilot study objectives. The starting dose will be 200 mg twice daily. Dosing will continue daily for 28 days, this being one cycle. There will be no protocol scheduled hiatus and daily dosing will be continuous unless there is unacceptable toxicity, disease progression, or death.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Participant will take 200 mg capsules or tablets orally twice daily. The participant will be instructed to swallow abemaciclib as a whole tablet and not to chew, crush or split capsules or tablets before swallowing. Participants should not ingest abemaciclib tablets if broken, cracked, or otherwise not intact. Doses should be taken at a approximately the same time every day, twice daily. Capsules or tablets can be taken orally with or without food. If the participant vomits or misses a dose of abemaciclib, the participant will be instructed to take the next dose at its scheduled time.
  Participants will also be provided with a diary and instructed to keep a twice daily record of the times they have taken their medications and any other events such as vomiting, diarrhea, etc.
  Other Names: Verzenio

SUMMARY:
The prognosis of patients with recurrent, late-stage inoperable, or progressed biliary tract carcinoma (BTC) is generally poor. The goal of this clinical study is to determine the effectiveness and safety of abemaciclib in patients with late-stage or progressed BTC that has failed one line of chemotherapy.

DETAILED DESCRIPTION:
Biliary Tract Carcinoma (BTC) is a leading cause of cancer-related mortality. The newly developed small molecule inhibitor of cyclin-dependent kinases (CDK4 and CDK6), abemaciclib, provides a new opportunity of treating patients with BTC. The goal of this clinical study is to determine the efficacy and safety of abemaciclib in patients with advanced or metastatic BTC that has progressed or intolerant to one or more lines of systemic therapy, or treatment-naïve subjects who either decline or being considered not a good candidate first-line systemic chemotherapy per the opinion of the treating physician.

The investigator's objectives for this study are as follows:

Primary Objectives:

• To estimate the objective response rate (ORR)

Secondary Objectives:

* To determine progression free survival (PFS)
* To determine the disease control rate (DCR)
* To determine the overall survival (OS) rate at 6 and 12 months
* To determine quality of life (QoL) using EORTC-QLQ-C30

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years at the time of informed consent.
2. Capable and willing to sign informed consent form prior to performing any protocol-related procedures.
3. Histologic or cytologic evidence of advanced or metastatic biliary tract cancer, including cholangiocarcinoma (intra-hepatic or extra-hepatic bile ducts), ampullary carcinoma, or gallbladder carcinoma.
4. Evidence of recurrent, locally advanced, unresectable, or metastatic disease.
5. Progressed following or intolerant to one or more lines of systemic therapy, or treatment-naïve subjects who either decline or being considered not a good candidate first-line systemic chemotherapy per the opinion of the treating physician
6. Per the opinion of the physician investigator, predicted life expectancy > 3 months.
7. Presence of at least 1 lesion that is measurable or evaluable using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
9. Per the opinion of the physician investigator, acute toxicities relating to any prior anticancer treatment have improved to Grade 1 or baseline. Exceptions include residual alopecia or Grade 2 peripheral neuropathy.
10. Ability to swallow capsules.
11. Adequate organ function as evidenced by the laboratory parameters noted in Section 3.0 Study Eligibility.
12. Women of childbearing potential (WOCP) defined as not surgically sterile (hysterectomy, tubal ligation, or oophorectomy), or at least 1 year postmenopausal, must have a negative serum pregnancy test before study drug administration on cycle 1 day 1.
13. WOCP must use a medically acceptable method of contraception and must agree to continue used of this method for the duration of the study and for 3 weeks after last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method.
14. Male, capable of producing offspring, must use a medical acceptable method of contraception and agree to continued use of this method for the duration of the study and for 3 weeks after last dose of study drug because of the possible effects on spermatogenesis. Acceptable methods of contraception include abstinence, WOCP partner's use of barrier method with spermicide, WOCP partner's use of an IUD known to have a failure rate of less than 1% per year, WOCP partner's use of steroidal contraceptive (oral, transdermal, implanted or injected) or WOCP partner is surgically sterile or at least 1 year post-menopausal. In addition, male subjects may not donate sperm for the duration of the study and for 30 days after last dose of study drug.
15. Must be willing and able to comply with the protocol, including adhering to study restrictions, remaining at the clinic as required during the study period, and willing to return to the clinic for the follow-up evaluation.
16. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy.
17. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
18. Completed last dose of myelosuppressive chemotherapy greater than 21 days prior to first dose of study drug.
19. Completed last dose of non-myelosuppressive biological or monoclonal antibody therapy greater than 14 days prior to first dose of study drug.

Exclusion Criteria:

1. Ongoing or active infection requiring systemic antibiotics.
2. Uncontrolled hypertension despite adequate therapy (systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 90 mm Hg found on 2 separate occasions separated by 1 week).
3. Diabetes mellitus and occurrence of more than 2 episodes of ketoacidosis in the 12 months prior to the first dose of study drug.
4. Active second malignancy other than curatively resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or other cancers treated with curative intent, and no known active disease in the 3 years prior to enrollment.
5. Primary brain tumor or brain metastases from another primary site.
6. Known history of human immunodeficiency virus (HIV).
7. Known active viral hepatitis B or viral hepatitis C.
8. History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Subjects with controlled atrial fibrillation for more than 30 days are permitted.
9. Congestive heart failure (New York Heart Association [NYHA] Class III or IV), or acute coronary syndromes within 6 months of enrollment.
10. Female subjects who are pregnant or breastfeeding.
11. Any other medical, psychiatric, or social condition, which in the opinion of the physician investigator, would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results. For example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy.
12. Use of an investigational drug within 1 month before the screening visit or currently participating in another investigational study.
13. Any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including extensive gastrointestinal surgery that involves removal of the entire stomach or most of the small intestine or large intestine, bariatric surgery, uncontrolled active Crohn's Disease or ulcerative colitis, or preexisting condition resulting in baseline Grade 2 or higher diarrhea). History of Whipple's procedure is permitted.
14. Known hypersensitivity to any of the components in abemaciclib including micro-crystalline cellulose 102, microcrystalline cellulose 101, lactose monohydrate, croscarmellose sodium, sodium stearyl fumarate, silicon dioxide. Color mixture ingredients-polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc, iron oxide yellow, and iron oxide red.
15. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Yee, MD, Ph.D, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This open-label pilot study aimed to evaluate the response and tolerability of abemaciclib (Verzenio) in patients with advanced biliary tract carcinoma. The primary purpose was to estimate the overall response rate in participants with locally advanced, unresectable, or metastatic biliary tract carcinoma who have failed first-line therapy.
Groups:
- Abemaciclib: Abemaciclib will be given as a single oral agent A sample size of 10 subjects is determined to be minimally sufficient for these pilot study objectives. The starting dose will be 200 mg twice daily. Dosing will continue daily for 28 days, this being one cycle. There will be no protocol scheduled hiatus and daily dosing will be continuous unless there is unacceptable toxicity, disease progression, or death.
  Abemaciclib: Participant will take 200 mg capsules or tablets orally twice daily. The participant will be instructed to swallow abemaciclib as a whole tablet and not to chew, crush or split capsules or tablets before swallowing. Participants should not ingest abemaciclib tablets if broken, cracked, or otherwise not intact. Doses should be taken at a approximately the same time every day, twice daily. Capsules or tablets can be taken orally with or without food. If the participant vomits or misses a dose of abemaciclib, the participant will be instructed to take the next dose at its scheduled time.
  Participants will also be provided with a diary and instructed to keep a twice daily record of the times they have taken their medications and any other events such as vomiting, diarrhea, etc.
Period: Overall Study
Arm/Group | Abemaciclib
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who were enrolled in the study before it was terminated. In this case, the study enrolled a total of 4 participants out of the planned 10.
Units Other Than Participants: tumor lesions
Arm/Group | Abemaciclib
Number analyzed (Participants) | 4
Number analyzed (tumor lesions) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: overall response rate (ORR) is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.The scale of ORR ranges from 0% to 100%, where 0% indicates no subjects achieved CR or PR, and 100% indicates all evaluable subjects achieved CR or PR.
Time Frame: no longer than 7 months
Population: No response data was collected as all participants were off treatment before the start of cycle 3, which is the earliest timepoint for ORR assessment.
Groups:
- Abemaciclib: Abemaciclib will be given as a single oral agent The starting dose will be 200 mg twice daily. Dosing will continue daily for 28 days, this being one cycle. There will be no protocol scheduled hiatus and daily dosing will be continuous unless there is unacceptable toxicity, disease progression, or death.
  Abemaciclib: Participant will take 200 mg capsules or tablets orally twice daily. The participant will be instructed to swallow abemaciclib as a whole tablet and not to chew, crush or split capsules or tablets before swallowing. Participants should not ingest abemaciclib tablets if broken, cracked, or otherwise not intact. Doses should be taken at a approximately the same time every day, twice daily. Capsules or tablets can be taken orally with or without food. If the participant vomits or misses a dose of abemaciclib, the participant will be instructed to take the next dose at its scheduled time.
  Participants will also be provided with a diary and instructed to keep a twice daily record of the times they have taken their medications and any other events such as vomiting, diarrhea, etc.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: the time interval from date of first dose of study drug to first documented disease progression or death from any cause, whichever occurs first. The PFS scale ranges from 0 days (for immediate progression or death) to the longest observed duration without progression or death.
Time Frame: through study completion, an average of 2 years
Population: Only two subjects with follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abemaciclib
Number analyzed (Participants) | 2
days | 110 (76)

3. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate (DCR) is defined as the proportion of subjects who achieve a Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. The scale of DCR ranges from 0% to 100%, where 0% indicates no subjects achieved CR, PR, or SD, and 100% indicates all evaluable subjects achieved disease control (CR, PR, or SD). Subjects who do not have sufficient data to determine response status are excluded from the denominator.
Time Frame: no longer than 7 months
Population: The number of subjects with CR, PR, or SD and the total number of subjects evaluable for response are detailed in the data tables.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate (OSR) is is typically reported as a percentage (%), representing the proportion of subjects who are alive at a specific time point after receiving the first dose of the study drug. The scale of Overall Survival Rate (OSR) ranges from 0% to 100%, where 0% indicates that none of the study participants survived for the specified period after the first dose of the study drug, and 100% indicates that all participants are alive at that time point. A higher OSR percentage suggests a greater proportion of subjects who have survived, reflecting the potential effectiveness of the treatment under investigation.
Time Frame: up to 6 months
Population: Two out of two evaluable subjects were alive at 6 months. No data available for 12-month survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 2
Participants | 2

5. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate (OSR) is is typically reported as a percentage (%), representing the proportion of subjects who are alive at a specific time point after receiving the first dose of the study drug. The scale of Overall Survival Rate (OSR) ranges from 0% to 100%, where 0% indicates that none of the study participants survived for the specified period after the first dose of the study drug, and 100% indicates that all participants are alive at that time point. A higher OSR percentage suggests a greater proportion of subjects who have survived, reflecting the potential effectiveness of the treatment under investigation. Overall Survival at 12 months is not available. Data were only collected up to 6 months.
Time Frame: up to 12 months
Population: No data available for 12-month survival.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life Score
Description: Quality of Life (QoL) will be assessed from the date of baseline and then every 4 weeks using the EORTC QLQ-C30. The QLQ-C30 comprises both multi-item scales and single-item measures, including a global health status/QoL scale, five functional scales, three multi-item symptom scales, and six single-item scales. For the multi-item scales, the raw score (RS) is calculated by taking the mean of the individual item scores. A linear transformation is then applied to standardize the raw score, resulting in a standardized score ranging from 0 to 100, where a score of 0 indicates the worst possible QoL and a score of 100 indicates the best possible QoL.
Time Frame: Prior to treatment with Abemaciclib (baseline)
Population: Four subjects completed EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abemaciclib
Number analyzed (Participants) | 4
score on a scale | 58.3 (37.9)

7. Secondary Outcome: Quality of Life Score
Description: as for outcome 6
Time Frame: Cycle 1 (28 days) treatment with Abemaciclib
Population: Three subjects completed EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abemaciclib
Number analyzed (Participants) | 3
score on a scale | 66.7 (30)

8. Secondary Outcome: Quality of Life Score
Description: as for outcome 6
Time Frame: Cycle 2 (56 days) treatment with Abemaciclib
Population: Three subjects completed EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abemaciclib
Number analyzed (Participants) | 3
score on a scale | 44.4 (25.5)

9. Secondary Outcome: Quality of Life Score
Description: as for outcome 6
Time Frame: Assessment at the end of treatment with Abemaciclib, approximately 60 days after starting treatment.
Population: Two subjects completed EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abemaciclib
Number analyzed (Participants) | 2
score on a scale | 29.2 (41.2)

ADVERSE EVENTS:
Time Frame: 1st subject: 1 month 2nd subject: 1 month 3rd subject: 2 months 4th subject: 2 months
Arm/Group | Abemaciclib
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=4)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 2 (5)
Abdominal Distension (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Chills (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Night sweat (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (General disorders) | 1 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (2)
BUN increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1)
Movements involuntary (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04003896/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04003896/ICF_001.pdf